CLINICAL TRIAL: NCT05383742
Title: A Phase II, Randomized, Open-Label Trial of a Six-Month Regimen of High-Dose Rifampicin, High-Dose Isoniazid, Linezolid, and Pyrazinamide Versus a Standard Nine-Month Regimen for the Treatment of Adults and Adolescents With Tuberculous Meningitis: Improved Management With Antimicrobial AGents Isoniazid rifampiciN LinEzolid for TBM (IMAGINE-TBM)
Brief Title: Trial of a Six-Month Regimen of High-Dose Rifampicin, High-Dose Isoniazid, Linezolid, and Pyrazinamide Versus a Standard Nine-Month Regimen for the Treatment of Adults and Adolescents With Tuberculous Meningitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5384
Record Dates: First submitted 2022-04-08; First posted 2022-05-20 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Tuberculous Meningitis
Keywords: Tuberculosis, meningeal; Tuberculosis; CNS Disease
MeSH Terms: conditions — Tuberculosis, Meningeal; Tuberculosis; Central Nervous System Diseases | interventions — Rifampin; Isoniazid; Linezolid; Pyrazinamide; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): RIF 35 mg/kg + INH 15 mg/kg + LZD 1200 mg + PZA 25 mg/kg for 2 weeks, followed by RIF 35 mg/kg + INH 10 mg/kg + LZD 1200 mg + PZA 25 mg/kg for 6 weeks, and then RIF 35 mg/kg and INH 10 mg/kg for 16 weeks, for a total of 24 weeks of study treatment.
  Interventions: Drug: Rifampicin (RIF); Drug: Isoniazid (INH); Drug: Linezolid (LZD); Drug: Pyrazinamide (PZA)
- Arm B (Active Comparator): WHO SOC: RIF 10 mg/kg + INH 5 mg/kg + ethambutol (EMB) 20 mg/kg + PZA 25 mg/kg for 8 weeks, followed by RIF 10 mg/kg and INH 5 mg/kg for 28 weeks, for a total of 36 weeks of study treatment. Up to 15 mg/kg or a maximum of 900 mg daily of oral RIF will be permitted in this arm at clinician's discretion.
  Interventions: Drug: Pyrazinamide (PZA); Drug: ethambutol (EMB); Drug: Rifampicin; Drug: Isoniazid

INTERVENTIONS:
Drug: Rifampicin (RIF) — Rifampicin 35 mg/kg
  Arms: Arm A
Drug: Isoniazid (INH) — Isoniazid 10 or15 mg/kg
  Arms: Arm A
Drug: Linezolid (LZD) — 1200 mg
  Arms: Arm A
Drug: Pyrazinamide (PZA) — 25 mg/kg
Drug: ethambutol (EMB) — 20 mg/kg
  Arms: Arm B
Drug: Rifampicin — 10 mg/kg
  Arms: Arm B
Drug: Isoniazid — 5 mg/kg
  Arms: Arm B

SUMMARY:
The purpose of this study is to compare a 6-month regimen of high-dose rifampicin (RIF), high-dose isoniazid (INH), linezolid (LZD), and pyrazinamide (PZA) versus the World Health Organization (WHO) standard of care (SOC) treatment for tuberculosis meningitis (TBM).

DETAILED DESCRIPTION:
Rationale: TBM is a devastating illness with high risk of mortality and severe neurologic morbidity. Although recent data suggest that significant dose increases in RIF may improve outcomes in TBM, mortality remains high, and enhanced treatment strategies are needed. In addition, limited data are available to guide treatment duration in adults with TBM. The overall goal of this Phase II, randomized, open-label trial is to assess the PK, safety, and longitudinal treatment outcomes of an optimized 6-month regimen of high-dose RIF, high-dose INH, LZD, and PZA to the WHO 9-month SOC regimen for the treatment of TBM.

Primary objective: To determine if a regimen of high-dose RIF, high-dose INH, LZD, and PZA improves functional outcomes measured by the modified Rankin Scale (mRS) at 48 weeks compared with WHO SOC for the treatment of TBM.

Design: Participants with definite, probable, or possible TBM will be randomized to one of the two study arms below and randomization will be stratified by HIV status and stage of disease as defined by the modified British Medical Research Council (BMRC) Classification TBM Grade.

Arm A: RIF 35 mg/kg + INH 15 mg/kg + LZD 1200 mg + PZA 25 mg/kg for 2 weeks, followed by RIF 35 mg/kg + INH 10 mg/kg + LZD 1200 mg + PZA 25 mg/kg for 6 weeks, and then RIF 35 mg/kg and INH 10 mg/kg for 16 weeks, for a total of 24 weeks of study treatment.

Arm B: WHO SOC: RIF 10 mg/kg + INH 5 mg/kg + EMB 20 mg/kg + PZA 25 mg/kg for 8 weeks, followed by RIF 10 mg/kg and INH 5 mg/kg for 28 weeks, for a total of 36 weeks of study treatment. Up to 15 mg/kg or a maximum of 900 mg daily of oral RIF will be permitted in this arm at clinician's discretion.

All participants in Arms A and B will receive pyridoxine, while receiving INH, and adjunctive corticosteroids according to BMRC TBM grade for at least 6 weeks.

All participants in Arms A and B will be followed from randomization to week 72.

Procedures: Study visits will include interval history, blood collection for laboratory testing, peripheral neuropathy screening, visual acuity, color vision, and contrast sensitivity visual testing to monitor for AEs. Lumbar puncture will be performed for assessments of CSF microbiology, LAM and other biomarkers. Optional collection and storage of blood and storage of remaining CSF for future testing will occur. Urine will be obtained for LAM assessment. Plasma and CSF PK assessments will be performed. Participants will undergo assessment of functional status with the mRS and WHO DAS 2.0. Participants will also be assessed with a neurocognitive battery and depression questionnaire (PHQ-9).

ELIGIBILITY:
Inclusion Criteria:

* Definite, probable, or possible TBM diagnosis wherein the participant is being committed to a full course of SOC anti-TB treatment for TBM in the setting of routine care. CSF, imaging, laboratory, and other results used to determine definite, probable, or possible TBM can be from testing performed as part of routine care, as long as obtained within 21 days prior to study entry
* Absence of HIV-1 infection, as documented by any licensed rapid HIV test or HIV-1 enzyme or chemiluminescence immunoassay (E/CIA) test kit, within 30 days prior to study entry, OR
* HIV-1 infection, documented by any licensed rapid HIV test or HIV-1 E/CIA test kit at any time prior to entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen or plasma HIV-1 RNA viral load. Two or more HIV-1 RNA viral loads of >1,000 copies/mL are also acceptable as documentation of HIV-1 infection, or documentation of HIV diagnosis in the medical record by a healthcare provider
* Documentation within 3 days prior to study entry of stage of disease using BMRC TBM grade.
* The following laboratory values obtained within 3 days prior to study entry:

  * Serum creatinine ≤1.8 times upper limit of normal (ULN)
  * Hemoglobin ≥8.0 g/dL for men, ≥7.5 g/dL for women
  * Absolute neutrophil count ≥600/mm3
  * Platelet count ≥60,000/mm3
  * Alanine aminotransferase (ALT) ≤3 x ULN
  * Total bilirubin ≤2 x ULN
* For participants of reproductive potential who have not been post-menopausal for at least 24 consecutive months (i.e., no menses within the preceding 24 months), or participants who have not undergone surgical sterilization, hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or tubal ligation, documentation of a serum or urine pregnancy test result (positive or negative; see protocol for test sensitivity requirement) within 21 days prior to study entry
* Participants with documentation of a positive pregnancy test will be consented using the consent form for pregnant participants.

Participants of reproductive potential with documentation of a negative pregnancy test must agree to use at least one acceptable form of contraception, or abstain from sexual activity that could lead to pregnancy while receiving study treatment and for 30 days after stopping study treatment.

Participants who are not of reproductive potential or whose partner(s) has documented azoospermia are not required to use contraception. Any statement of self-reported sterility or that of the partner's must be entered in the source documents

* Ability and willingness of participant or parent or legally authorized representative (for adolescents or participants unable to provide consent) to provide informed consent/assent
* Ability to comply with the protocol requirements in the opinion of the site investigator

Exclusion Criteria:

* More than 14 cumulative days of first-line TB medications, including but not limited to INH, RIF, EMB, and PZA, received within 90 days prior to study entry
* Known current or previous drug resistant TB infection (i.e., resistance to one or more first-line TB medications, including but not limited to INH, RIF, EMB, LZD and PZA)
* Known allergy/sensitivity or any hypersensitivity to components of study TB drugs (INH, RIF, LZD, PZA, and EMB) or their formulation
* For participants who are able to undergo the Brief Peripheral Neuropathy Screen (BPNS) within 21 days prior to study entry, Grade 3 subjective peripheral neuropathy score on the BPNS AND EITHER vibratory loss OR absent ankle jerks
* Expected concomitant use or use up to 21 days prior to study entry of monoamine oxidase inhibitors or selective serotonin reuptake inhibitors, or concomitant use of any other drug with significant interaction with the study drugs (See protocol)
* For participants with HIV who are ART-naïve or who are not regularly taking ART, planned initiation or reinitiation of ART during screening or during the first 4 weeks after initiation of TB therapy
* For participants with HIV and on ART that includes a protease inhibitor, nevirapine, or other prohibited ART (see protocol), contraindication to switching to an acceptable alternative regimen (e.g., efavirenz, high-dose raltegravir or dolutegravir with nucleoside reverse transcriptase inhibitors, as per local SOC) prior to randomization. TB treatment, including study drugs, should be started as soon as possible
* Contraindication to LP at discretion of treating clinician (e.g., unequal pressures between intracranial compartments due to mass lesion, non-communicating hydrocephalus)
* Positive cryptococcal antigen, gram stain, bacterial culture, or other test result obtained from a CSF specimen collected within 21 days prior to entry as part of routine care indicating CNS infection with a pathogen other than Mtb (e.g., cryptococcal meningitis, bacterial meningitis).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (6-death, 5-severe disability, 4-moderately severe disability, 3-moderate disability, 2-slight disability, 1-no significant disability, 0-no symptoms) | At 48 weeks

SECONDARY OUTCOMES:
Modified Rankin Scale (all 7 levels) | At 0, 12, 24, 36, 48 and 72 weeks
Modified Rankin Scale using collapsed categories: mRS (0 or 1), (2 or 3), (4 or 5), (6) | At 12, 24, 36, 48 and 72 weeks
Modified Rankin Scale 5 or 6 | At 12, 24, 36, 48 and 72 weeks
Time to death through 48 and 72 weeks | At weeks 48 and 72
Proportion of participants with Grade 3 or higher AEs | At 4, 8 and 24 weeks
Proportion of participants with a serious adverse event (SAE) | At 4, 8 and 24 weeks
Proportion of participants with study treatment discontinuations | At 4, 8 and 24 weeks
Proportion of participants who complete study treatments | At 185 and 278 days
Proportion of participants with TBM IRIS or paradoxical worsening | At 48 weeks
Wechsler Adult Intelligence Scale Digit Symbol | At 24 and 48 weeks
  Neurocognitive battery performance
Color Trails 1 | At 24 and 48 weeks
  Neurocognitive battery performance
Color Trails 2 | At 24 and 48 weeks
  Neurocognitive battery performance
Category Fluency | At 24 and 48 weeks
  Neurocognitive battery performance
Hopkins Verbal Learning Test-Revised | At 24 and 48 weeks
  Neurocognitive battery performance
Grooved Pegboard Bilateral | At 24 and 48 weeks
  Neurocognitive battery performance
Finger-tapping Bilateral | At 24 and 48 weeks
  Neurocognitive battery performance
Patient Health Questionnaire (PHQ-9) total score | At 24, 48, and 72 weeks
WHO DAS score | At 24, 48, and 72 weeks
Change in BMRC TBM grade at week 1 | At 1 week
Time to coma clearance | At 4 weeks
Time to new neurological event | At 48 weeks

OTHER OUTCOMES:
Proportion of participants with recurrence | At 36 and 48 weeks
Positive or negative CSF Xpert Ultra | At screening, Day 3 and week 2 or week 6 or week 8
Positive or negative CSF and urine LAM | At screening, Day 3 and week 2 or week 6 or week 8
Functional outcomes and mortality in definite TBM patients | At 72 weeks
Association of TBM host immune signatures and functional outcomes and treatment response | At 72 weeks
Change in sterilization of CSF culture | At Weeks 2 and 6-8
Change in CSF white blood cell count | At Weeks 2 and 6-8
Change in CSF glucose | At Weeks 2 and 6-8
Change in CSF blood glucose ratio | At Weeks 2 and 6-8
Change in CSF protein | At Weeks 2 and 6-8

CONTACTS AND LOCATIONS:
Locations (18):
- Brazil (2):
  - Hospital Nossa Senhora da Conceicao CRS (Site ID: 12201), Porto Alegre
  - Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS (Site ID: 12101), Rio de Janeiro
- Byramjee Jeejeebhoy Government Medical College (BJMC) CRS (Site ID: 31441), Pune, India
- Kenya (2):
  - Moi University Clinical Research Center (MUCRC) CRS (Site ID: 12601), Eldoret
  - Kenya Medical Research Institute/Walter Reed Project Clinical Research Center (KEMRI/WRP) CRS (Site ID: 12501), Kericho
- Malawi CRS (Site ID: 12001), Lilongwe, Malawi
- Nutrición-Mexico CRS (Site ID: 32078), Mexico City, Mexico
- Peru (2):
  - Socios en Salud Sucursal Peru CRS (Site ID: 31985), Lima
  - Barranco CRS (Site ID:11301), Lima
- TB HIV Innovations and Clinical Research Foundation Corp (Site ID: 31981), Cavite, Philippines
- South Africa (2):
  - Durban International CRS (Site ID:11201), Durban
  - University of the Witwatersrand Helen Joseph (WITS HJH) CRS (Site ID: 11101), Johannesburg
- Kilimanjaro Christian Medical Centre (KCMC) (Site ID: 5118), Moshi, Tanzania
- Thailand (3):
  - Siriraj Hospital, Mahidol University NICHD CRS (Site ID: 5115), Bangkok, Bangkoknoi
  - Thai Red Cross AIDS Research Centre (TRC-ARC) CRS (Site ID: 31802), Bangkok, Pathumwan
  - Chiangrai Prachanukroh Hospital NICHD CRS (Site ID: 5116), Chiang Mai
- National Lung Hospital CRS (Site ID: 32483), Vĩnh Phúc, Hanoi, Vietnam
- Milton Park CRS (Site ID: 30313), Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (ACTG) by NIH
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the ACTG.
  * For what types of analyses? To achieve aims in the proposal approved by the ACTG.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the ACTG "Data Request" form at: https://submit.mis.s-3.net/. Researchers of approved proposals will need to sign an ACTG Data Use Agreement before receiving the data